CLINICAL TRIAL: NCT01709305
Title: A Multicenter, Randomized, Active-Controlled, Open-label Clinical Trial to Evaluate the Safety and Efficacy of Glimepiride, Gliclazide, Repaglinide or Acarbose as a Third OAHA on Top of Sitagliptin+Metformin Combination Therapy in Chinese Patients With Type 2 Diabetes Mellitus
Brief Title: A Study of the Safety and Efficacy of Glimepiride, Gliclazide, Repaglinide or Acarbose When Added to Sitagliptin + Metformin Combination Therapy in Chinese Participants With Diabetes (MK-0431-313)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-313
Record Dates: First submitted 2012-10-16; First posted 2012-10-18 (Estimated); Results first posted 2016-05-11 (Estimated); Last update posted 2018-08-21 (Actual); Status verified 2018-07

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Metformin; Sitagliptin Phosphate; Acarbose; repaglinide; glimepiride; Gliclazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Metformin + Sitagliptin + Glimepiride (Active Comparator): During Phase 2, participants receive up to 6 mg glimepiride daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44).
  Interventions: Drug: Metformin; Drug: Sitagliptin; Drug: Glimepiride
- Metformin + Sitagliptin + Repaglinide (Experimental): During Phase 2, participants receive up to 16 mg repaglinide daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44).
  Interventions: Drug: Metformin; Drug: Sitagliptin; Drug: Repaglinide
- Metformin + Sitagliptin + Acarbose (Experimental): During Phase 2, participants receive 50-100 mg acarbose three times daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44).
  Interventions: Drug: Metformin; Drug: Sitagliptin; Drug: Acarbose
- Metformin + Sitagliptin + Gliclazide (Experimental): During Phase 2, participants receive 30-120 mg gliclazide daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44).
  Interventions: Drug: Metformin; Drug: Sitagliptin; Drug: Gliclazide

INTERVENTIONS:
Drug: Metformin — Metformin, 500 mg or 850 mg oral tablets, twice or three times a day (BID or TID) for a total dose of at least 1500 mg daily; administered with food.
  Other Names: Fortamet®; Glucophage®; Glucophage® XR; Glumetza®; Riomet®; Metgluco®; Glycoran®
Drug: Sitagliptin — Sitagliptin, 100 mg oral tablet, once daily (QD); administered with or without food
  Other Names: Januvia®; Tesavel®; Xelevia®; Ristaben®
Drug: Acarbose — Acarbose, 50 mg oral tablets, TID (150 mg total daily dose); administered with the first bite of each main meal.
  Other Names: Precose®; Glucobay™
  Arms: Metformin + Sitagliptin + Acarbose
Drug: Repaglinide — Repaglinide, 0.5 mg and/or 1 mg oral tablets, TID (up to 16 mg daily); administered within 30 minutes of each meal.
  Other Names: Prandin®; Fulaidi™
  Arms: Metformin + Sitagliptin + Repaglinide
Drug: Glimepiride — Glimepiride, 1 mg and/or 2 mg oral tablets, QD (up to 6 mg daily); administered before the first main meal of the day
  Other Names: Amaryl®; Glimy
  Arms: Metformin + Sitagliptin + Glimepiride
Drug: Gliclazide — Gliclazide, 30 mg oral tablets, QD or BID (30 mg to 120 mg total daily dose); administered with meal.
  Other Names: Diamicron MR™
  Arms: Metformin + Sitagliptin + Gliclazide

SUMMARY:
To assess the effect of adding acarbose or repaglinide or gliclazide to sitagliptin plus metformin, compared to adding glimepiride, on glycemic improvements in Type 2 Diabetes Mellitus (T2DM) participants who require the addition of a third oral anti-hyperglycemic agent (OAHA) according to China Guideline for Type 2 Diabetes. The three co-primary hypotheses are that after 24 weeks of treatment in phase 2, the mean change from baseline in hemoglobin A1c (A1c) in participants receiving either (1)acarbose or (2)repaglinide or (3)gliclazide added to sitagliptin and metformin combination is non-inferior to that of participants receiving glimepiride added to sitagliptin and metformin combination. The study would be declared successful if at least one of the three primary hypotheses was met.

DETAILED DESCRIPTION:
Participants coming on study will be stabilized to a standardized metformin dose: this may take about 10 weeks, and then combination therapy with metformin + sitagliptin will begin during Phase 1 (Week 0 through Week 20). If a participant has already been on a stabilized metformin dose, they will start immediately on combination therapy with metformin + sitagliptin for 20 weeks (Phase 1).

In Phase 2, participants who have failed to achieve adequate glycemic control (A1c ≥ 7% and ≤ 10% at Week 16 and fasting finger stick glucose ≥130 mg/dL and ≤280 mg/dL at Week 20) will be randomized to receive add-on therapy with glimepiride, repaglinide, acarbose, or gliclazide for 24 weeks (Week 20 through Week 44).

ELIGIBILITY:
Inclusion Criteria:

* Has Type 2 Diabetes Mellitus;
* Agrees to use an effective method of contraception or must not otherwise be at risk of becoming pregnant (female participants).

Exclusion Criteria:

* Has a history of type 1 diabetes mellitus or a history of ketoacidosis;
* Has been treated with insulin, a dipeptidyl peptidase 4 (DPP-4) inhibitor, a Glucagon-like peptide-1 (GLP-1) mimetic or analogue before;
* Is on a weight loss program (not in maintenance phase), has started a weight loss medication, or has undergone bariatric surgery within 12 months;
* Has undergone a surgical procedure within 4 weeks;
* Has had new or worsening signs or symptoms of coronary heart disease or congestive heart failure within past 3 months, or has acute coronary syndrome, coronary artery intervention, or stroke or transient ischemic neurological disorder;
* Has a medical history of active liver disease, including chronic active hepatitis B or C, primary biliary cirrhosis, or symptomatic gallbladder disease;
* Has poorly controlled hypertension;
* Has severe peripheral vascular disease;
* Has human immunodeficiency virus (HIV);
* Has had a clinically important hematological disorder;
* Routinely consumes >2 alcoholic drinks per day or >14 alcoholic drinks per week, or engages in binge drinking;
* Has a history of intolerance or hypersensitivity or any contraindication to study medications (including sitagliptin, metformin, glimepiride, repaglinide, acarbose or gliclazide) based upon the Chinese label;
* Is on or likely to require treatment with ≥2 consecutive weeks or repeated courses of pharmacologic doses of corticosteroids (other than inhaled, nasal, or topical corticosteroids);
* Is pregnant or breast feeding or is expecting to conceive or donate eggs during the study, including 14 days following the last dose of study drug (female participants).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5570 (Actual)
Dates: Start 2012-11-08 (Actual); Primary Completion 2015-04-17 (Actual); Study Completion 2015-04-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Xu W, Mu Y, Zhao J, Zhu D, Ji Q, Zhou Z, Yao B, Mao A, Engel SS, Zhao B, Bi Y, Zeng L, Ran X, Lu J, Ji L, Yang W, Jia W, Weng J. Efficacy and safety of metformin and sitagliptin based triple antihyperglycemic therapy (STRATEGY): a multicenter, randomized, controlled, non-inferiority clinical trial. Sci China Life Sci. 2017 Mar;60(3):225-238. doi: 10.1007/s11427-016-0409-7. Epub 2017 Feb 7. PMID 28271251

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult Chinese participants (≥18 and ≤75 years of age) with a diagnosis of Type 2 Diabetes Mellitus (T2DM) and inadequate glycemic control were selected to participate in this study.
Pre-assignment Details: There were 2344 participants who achieved A1C<7% in Phase 1; they completed Phase 1 and did not enter Phase 2. Of the remaining 2589 participants, 377 participants did not meet randomization criteria to enter Phase 2.
Groups:
- Phase 1: Sitagliptin + Metformin: During Phase 1, participants received sitagliptin 100 mg + metformin (Week 0 through Week 20). There were 5570 participants enrolled in Phase 1.
- Phase 2: Metformin + Sitagliptin + Glimepiride: During Phase 2, participants received up to 6 mg glimepiride daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44). There were 552 participants randomized to this arm in Phase 2.
- Phase 2: Metformin + Sitagliptin + Repaglinide: During Phase 2, participants received up to 16 mg repaglinide daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44). There were 550 participants randomized to this arm in Phase 2.
- Phase 2: Metformin + Sitagliptin + Acarbose: During Phase 2, participants received 50-100 mg acarbose three times daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44). There were 556 participants randomized to this arm in Phase 2.
- Phase 2: Metformin + Sitagliptin + Gliclazide: During Phase 2, participants received 30-120 mg gliclazide daily as an add-on to metformin + sitagliptin combinatino therapy for 24 weeks (Week 20 through Week 44). There were 554 participants randomized to this arm in Phase 2.
Period: Phase 1
Arm/Group | Phase 1: Sitagliptin + Metformin | Phase 2: Metformin + Sitagliptin + Glimepiride | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Gliclazide
Started | 5570 | 0 | 0 | 0 | 0
Completed | 4933 | 0 | 0 | 0 | 0
Not Completed | 637 | 0 | 0 | 0 | 0
Not completed — Clinical Adverse Event | 80 | 0 | 0 | 0 | 0
Not completed — Death | 2 | 0 | 0 | 0 | 0
Not completed — Hyperglycemia (lack of efficacy) | 13 | 0 | 0 | 0 | 0
Not completed — Laboratory Adverse Event | 16 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 147 | 0 | 0 | 0 | 0
Not completed — Travel, moving, etc. | 30 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 13 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 118 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 218 | 0 | 0 | 0 | 0
Period: Phase 2
Arm/Group | Phase 1: Sitagliptin + Metformin | Phase 2: Metformin + Sitagliptin + Glimepiride | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Gliclazide
Started | 0 | 552 | 550 | 556 | 554
Completed | 0 | 500 | 505 | 508 | 507
Not Completed | 0 | 52 | 45 | 48 | 47
Not completed — Clinical Adverse Event | 0 | 10 | 10 | 6 | 11
Not completed — Death | 0 | 0 | 1 | 0 | 0
Not completed — Hyperglycemia (lack of efficacy) | 0 | 0 | 0 | 0 | 2
Not completed — Laboratory Adverse Event | 0 | 1 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 10 | 6 | 9 | 5
Not completed — Travel, moving, etc. | 0 | 2 | 3 | 3 | 5
Not completed — Physician Decision | 0 | 2 | 0 | 1 | 2
Not completed — Protocol Violation | 0 | 19 | 19 | 13 | 9
Not completed — Withdrawal by Subject | 0 | 8 | 6 | 15 | 12

BASELINE CHARACTERISTICS:
Population: This population includes all participants who enrolled in Phase 1 and were GCP compliant.
Groups:
- Overall Study: During Phase 1, participants received sitagliptin 100 mg + metformin (Week 0 through Week 20).
Arm/Group | Overall Study
Number analyzed (Participants) | 5535
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.1 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2240
  Male | 3295

OUTCOME MEASURES:

1. Primary Outcome: Change From Phase 2 Baseline to Week 44 in Hemoglobin A1c (HbA1c) Levels (Phase 2)
Description: HbA1c is blood marker used to report average blood glucose levels over prolonged periods of time and is reported as a percentage (%). Change from baseline reflects the Week 44 A1C minus baseline A1C. Baseline is defined as Visit 6/Week 20. If this measurement was unavailable, the Week 16 value was used. Change from baseline was based on the constrained longitudinal data analysis (cLDA) model including all available measurements from baseline through the last visit. The terms in the cLDA model include treatment, time in weeks (categorical), regions, and treatment-by-time interaction.
Time Frame: Phase 2 Baseline (Week 20) and Week 44
Population: Per-Protocol (PP) population - excluded those participants who were identified as protocol violators and those who were non-compliant with Good Clinical Practice (GCP) requirements.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Groups:
- Phase 2: Metformin + Sitagliptin + Glimepiride: During Phase 2, participants received up to 6 mg glimepiride daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44).
- Phase 2: Metformin + Sitagliptin + Repaglinide: During Phase 2, participants received up to 16 mg repaglinide daily as an add-on to metfomin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44).
- Phase 2: Metformin + Sitagliptin + Acarbose: During Phase 2, participants received 50-100 mg acarbose three times daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44).
- Phase 2: Metformin + Sitagliptin + Gliclazide: During Phase 2, participants received 30-120 mg gliclazide daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44).
Arm/Group | Phase 2: Metformin + Sitagliptin + Glimepiride | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Gliclazide
Number analyzed (Participants) | 414 | 418 | 472 | 418
Percent | -0.65 (0.84) [-0.73 to -0.57] | -0.62 (0.84) [-0.69 to -0.54] | -0.46 (0.83) [-0.53 to -0.38] | -0.69 (0.90) [-0.77 to -0.61]
Statistical Analysis 1: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Acarbose; Pairwise Comparison; Test type: Non-Inferiority or Equivalence — Non-inferiority criterion are met when the upper limit of the two-sided 98.34% CI for the difference in LS means is less than or equal to the pre-specified non-inferiority margin of 0.3%; Difference in LS Means = 0.19, 98.34% CI 2-sided [0.02 to 0.36]
Statistical Analysis 2: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Repaglinide; Pairwise Comparison; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in LS Means = 0.03, 98.34% CI 2-sided [-0.15 to 0.21]
Statistical Analysis 3: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Gliclazide; Pairwise Comparison; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Difference in LS Means = -0.05, 98.34% CI 2-sided [-0.23 to 0.14]

2. Secondary Outcome: Change From Phase 2 Baseline to Week 44 in Participant Body Weight (Phase 2)
Description: Change from baseline in body weight in Phase 2 was reported. Change from baseline reflects the Week 44 body weight minus baseline body weight. Baseline is defined as Visit 6/Week 20. If this measurement was unavailable, the Week 16 value was used.
Time Frame: Phase 2 Baseline (Week 20), Week 44
Population: All Participants as Treated (APaT) - all randomized participants who received at least one (1) dose of study treatment and were compliant with GCP requirements.
Measure: Mean (Standard Deviation); unit: kg
Groups:
- Phase 2: Metformin + Sitagliptin + Glimepiride: During Phase 2, participants received up to 6 mg glimepiride daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44). There were 501 participants that contributed to the week 44 analysis.
- Phase 2: Metformin + Sitagliptin + Repaglinide: During Phase 2, participants received up to 16 mg repaglinide daily as an add-on to metfomin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44). There were 502 participants that contributed to the week 44 analysis.
- Phase 2: Metformin + Sitagliptin + Acarbose: During Phase 2, participants received 50-100 mg acarbose three times daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44). There were 551 participants that contributed to the week 44 analysis.
- Phase 2: Metformin + Sitagliptin + Gliclazide: During Phase 2, participants received 30-120 mg gliclazide daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44). There were 550 participants that contributed to the week 44 analysis.
Arm/Group | Phase 2: Metformin + Sitagliptin + Glimepiride | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Gliclazide
Number analyzed (Participants) | 501 | 502 | 509 | 506
kg | 0.4 (2.6) | 0.2 (2.5) | -0.9 (2.5) | 0.2 (2.4)

3. Secondary Outcome: Percentage of Participants With Hypoglycemia Events (Phase 2)
Description: Hypoglycemia events represent epidsodes symptomatic of hypoglycemia (e.g., weakness, dizziness, shakiness, increased sweating, palpitations, or confusion) and/or finger stick glucose values of ≤70 mg/dL (3.9 mmol/L). The percentage of participants with hypoglycemia events was reported.
Time Frame: From Week 20 through Week 44
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: Metformin + Sitagliptin + Glimepiride | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Gliclazide
Number analyzed (Participants) | 549 | 545 | 551 | 550
Percentage of Participants | 8.9 | 6.1 | 0.5 | 3.6
Statistical Analysis 1: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Acarbose; Difference in % vs. Glimepiride; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen; Estimate = -8.4, 95% CI 2-sided [-11.1 to -6.1]
Statistical Analysis 2: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Repaglinide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.072, Miettinen & Nurminen; Estimate = -2.9, 95% CI 2-sided [-6.1 to 0.3]
Statistical Analysis 3: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Gliclazide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p < 0.001, Miettinen & Nurminen; Estimate = -5.3, 95% CI 2-sided [-8.3 to -2.5]

4. Secondary Outcome: Percentage of Participants With a Gastrointestinal (GI) AE of Nausea (Phase 2)
Description: The percentage of participants with a GI AE of "nausea" was reported.
Time Frame: From Week 20 through Week 44
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: Metformin + Sitagliptin + Glimepiride | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Gliclazide
Number analyzed (Participants) | 549 | 545 | 551 | 550
Percentage of Participants | 0 | 0 | 0.4 | 0.2
Statistical Analysis 1: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Acarbose; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.158, Miettinen & Nurminen; Estimate = 0.4, 95% CI 2-sided [-0.3 to 1.3]
Statistical Analysis 2: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Repaglinide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p > 0.999, Miettinen & Nurminen; Estimate = 0.0, 95% CI 2-sided [-0.7 to 0.7]
Statistical Analysis 3: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Gliclazide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.318, Miettinen & Nurminen; Estimate = 0.2, 95% CI 2-sided [-0.5 to 1.0]

5. Secondary Outcome: Percentage of Participants With a GI AE of Vomiting (Phase 2)
Description: The percentage of participants with a GI AE of "vomiting" was reported.
Time Frame: From Week 20 through Week 44
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: Metformin + Sitagliptin + Glimepiride | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Gliclazide
Number analyzed (Participants) | 549 | 545 | 551 | 550
Percentage of Participants | 0.2 | 0 | 0.2 | 0.2
Statistical Analysis 1: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Acarbose; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.998, Miettinen & Nurminen; Estimate = -0.0, 95% CI 2-sided [-0.9 to 0.9]
Statistical Analysis 2: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Repaglinide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.319, Miettinen & Nurminen; Estimate = -0.2, 95% CI 2-sided [-1.0 to 0.5]
Statistical Analysis 3: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Gliclazide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.999, Miettinen & Nurminen; Estimate = -0.0, 95% CI 2-sided [-0.9 to 0.9]

6. Secondary Outcome: Percentage of Participants With a GI AE of Diarrhea (Phase 2)
Description: The percentage of participants with a GI AE of "diarrhea" was reported.
Time Frame: From Week 20 through Week 44
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: Metformin + Sitagliptin + Glimepiride | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Gliclazide
Number analyzed (Participants) | 549 | 545 | 551 | 550
Percentage of Participants | 0.5 | 0.4 | 0.4 | 0.9
Statistical Analysis 1: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Acarbose; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.651, Miettinen & Nurminen; Estimate = -0.2, 95% CI 2-sided [-1.3 to 0.8]
Statistical Analysis 2: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Repaglinide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.660, Miettinen & Nurminen; Estimate = -0.2, 95% CI 2-sided [-1.3 to 0.8]
Statistical Analysis 3: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Gliclazide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.480, Miettinen & Nurminen; Estimate = 0.4, 95% CI 2-sided [-0.8 to 1.6]

7. Secondary Outcome: Percentage of Participants With a GI AE of Abdominal Pain (Phase 2)
Description: The percentage of participants with a GI AE of "abdominal pain" was reported.
Time Frame: From Week 20 through Week 44
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Phase 2: Metformin + Sitagliptin + Glimepiride | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Gliclazide
Number analyzed (Participants) | 549 | 545 | 551 | 550
Percentage of Participants | 0 | 0 | 0.4 | 0.2
Statistical Analysis 1: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Acarbose; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.158, Miettinen & Nurminen; Estimate = 0.4, 95% CI 2-sided [-0.3 to 1.3]
Statistical Analysis 2: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Repaglinide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p > 0.999, Miettinen & Nurminen; Estimate = 0.0, 95% CI 2-sided [-0.7 to 0.7]
Statistical Analysis 3: Comparison: Phase 2: Metformin + Sitagliptin + Glimepiride vs Phase 2: Metformin + Sitagliptin + Gliclazide; Difference in % vs. Glimepiride; Test type: Superiority or Other; p = 0.318, Miettinen & Nurminen; Estimate = 0.2, 95% CI 2-sided [-0.5 to 1.0]

ADVERSE EVENTS:
Time Frame: Up to 46 Weeks
Description: All Participants as Treated (APaT) - all participants enrolled (Phase 1) or randomized (Phase 2) who received at least one dose of study treatment and complied with GCP requirements. Participants were included in the treatment group corresponding to the study treatment they actually received.
Groups:
- Phase 1: Sitagliptin + Metformin: During Phase 1, participants received sitagliptin 100 mg + metformin for 20 weeks (Week 0 through Week 20).
- Phase 2: Metformin + Sitagliptin + Repaglinide: During Phase 2, participants received up to 16 mg repaglinide daily as an add-on to metformin + sitagliptin combination therapy for 24 weeks (Week 20 through Week 44).
Arm/Group | Phase 1: Sitagliptin + Metformin | Phase 2: Metformin + Sitagliptin + Acarbose | Phase 2: Metformin + Sitagliptin + Repaglinide | Phase 2: Metformin + Sitagliptin + Gliclazide | Phase 2: Metformin + Sitagliptin + Glimepiride
Serious Adverse Events (participants affected / at risk) | 63/5527 | 11/551 | 9/545 | 10/550 | 8/549
Other Adverse Events (participants affected / at risk) | 66/5527 | 3/551 | 33/545 | 20/550 | 48/549
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Sitagliptin + Metformin (N=5527) | Phase 2: Metformin + Sitagliptin + Acarbose (N=551) | Phase 2: Metformin + Sitagliptin + Repaglinide (N=545) | Phase 2: Metformin + Sitagliptin + Gliclazide (N=550) | Phase 2: Metformin + Sitagliptin + Glimepiride (N=549)
Angina Pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina Unstable (Cardiac disorders) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis Coronary Artery (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Retinopathy (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Entropion (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Optic Ischaemic Neuropathy (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pterygium (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric Polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Large Intestine Polyp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sudden Death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Hepatopathy (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic Function Abnormal (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anal Abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Epididymitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis Media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spermatic Cord Funiculitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vestibular Neuronitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar Vertebral Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Meniscus Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Road Traffic Accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetes Mellitus Inadequate Control (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Diabetic Ketoacidosis (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Brain Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gallbladder Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian Adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatic Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroid Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid Arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral Haematoma (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral Infarction (Nervous system disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Lacunar Infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myasthenia Gravis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus Bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal Colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diabetic Foot (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug Eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incisional Drainage (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Interventional Procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Essential Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Varicose Ulceration (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute Myocardial Infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Duodenal Ulcer Haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis Acute (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vascular Stent Occlusion (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Liver Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gouty Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelodysplastic Syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tongue Neoplasm Malignant Stage Unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic Neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vertebrobasilar Insufficiency (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nephrotic Syndrome (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Artery Stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Sitagliptin + Metformin (N=5527) | Phase 2: Metformin + Sitagliptin + Acarbose (N=551) | Phase 2: Metformin + Sitagliptin + Repaglinide (N=545) | Phase 2: Metformin + Sitagliptin + Gliclazide (N=550) | Phase 2: Metformin + Sitagliptin + Glimepiride (N=549)
Hypoglycemia (Metabolism and nutrition disorders) | 66 (84) | 3 (5) | 33 (51) | 20 (35) | 48 (72)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the study without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.